CLINICAL TRIAL: NCT06251284
Title: Expectation Effects on Emotional Processing in Late Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Stefanie Brassen, Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PV7141
Record Dates: First submitted 2024-01-24; First posted 2024-02-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Expectation Effects on Emotional Processing in Late Life
Keywords: Positive expectation; fMRI; Attentional mechanisms; Cognitive control; Aging

STUDY DESIGN:
Intervention Model Description: A cross-over design will be employed by giving a saline nasal spray introduced either as oxytocin or as saline.
Who Masked: Participant
Masking Description: Participants will be blinded to the real substance (saline nasal spray).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo - Control (Experimental): Participants in this group receive sham oxytocin on the first study day.
  Interventions: Other: Saline nasal spray
- Control - Placebo (Experimental): Participants in this group receive sham oxytocin on the second study day
  Interventions: Other: Saline nasal spray

INTERVENTIONS:
Other: Saline nasal spray — A saline nasal spray will be introduced as saline on the first day (no induced expectations) and as oxytocin on the second day (induced positive expectations)

SUMMARY:
Understanding the mechanisms of expectation effects in the affective system is vital, given high placebo rates in antidepressants. Evidence has consistently confirmed that expectations can influence our emotional experience. Recently, a crucial role of prefrontal top-down regulation and cognitive capacity was shown in verbally instructed expectation effects within the affective system.

Empirical findings systematically point to a positivity effect in emotionally healthy aging, linked to prefrontal functioning. It is unclear whether the effects and mechanisms of positive expectations on emotional processing might also change throughout the lifespan. Hence, the investigators' goal is to explore the neurobehavioral mechanisms underlying positive expectation effects in healthy aging. Healthy older adults (N=55; 50% female) will be invited to a cross-over (positive expectation vs. no expectations induced) fMRI experiment during which they will perform an emotional interference task that manipulates cognitive resources. The investigators hypothesize that older adults demonstrate a resource-dependent positivity effect and that this effect will be further enhanced through the induction of positive expectations. Additionally, it is expected that these result are related to participants' general cognitive control ability and to be reflected on the corresponding neural correlates in prefrontal-limbic networks.

DETAILED DESCRIPTION:
Understanding the mechanisms of expectation effects on mood states and emotion processing can be crucial to develop depression treatment strategies. Evidence has related positive expectations to a perception bias towards positive information and changes in neural networks of affective processing. In a recent study conducted by our group, the investigators showed that verbally instructed positive expectations in healthy young adults improved subjective mood, reduced distractibility by aversive stimuli and activated top-down regulation processes in neural networks of emotion regulation. Moreover, these findings were related to cognitive control ability, mediated by prefrontal-parietal networks involved in attentional orienting. Together, these results emphasize the crucial role of top-down control regulation processes and cognitive capacity in verbally instructed expectation effects within the affective system. Additionally, evidence has frequently pointed to a positivity effect in emotionally healthy aging, linked to prefrontal functioning. This suggests that older adults tend to focus more on positive information compared to younger adults. It is unclear whether the effects and mechanisms of positive expectations on emotional processing change throughout the lifespan, assuming age-related alterations might affect neural networks responsible for emotional regulation and cognitive control in expectation effects. Therefore, the aim of this study is to investigate whether older adults also benefit from positive expectations and which neurobehavioral mechanisms and brain areas are related to this phenomenon.

Applying our previously established experimental setup, in this study, the investigators will invite 55 older healthy adults to participate in two fMRI sessions. During an initial screening, participants will complete demographic and psychometric questionnaires (Beck Depression Inventory (BDI) and previous experience with oxytocin). In addition, cognitive healthiness will be ensured via the Montreal Cognitive Assessment (MoCA) and participants will perform a visual search task to assess cognitive control ability (Singleton Task).

On two study days (separated by ~ 1 week), participants will undergo fMRI scanning. Before scanning, they will receive a saline nasal spray, introduced as oxytocin ("oxytocin" condition) or saline ("control" condition) in a counterbalanced cross-over design. Positive expectations about oxytocin will be induced by a custom 5-minute video documentary. After the video, participants will be told whether they are in the "oxytocin" or "control" condition and then self-administer the nasal-spray. Participants will report their expectations through a 11-point-scale (0 for no expected mood enhancement and 10 for large expected mood enhancement, GEEE) as well as mood state using a visual analogue scale (VAS) before the application of the nasal spray, during and after the fMRI measure. In the scanner, they will perform an emotion-interference task. The task is a modified spatial cueing paradigm, established in our lab. Participants will have to respond to left- or right- sided dots that are preceded by a spatially informative cue (arrow pointing to the side where the dot is most likely to appear) or uninformative cue (doubled arrow pointing to both sides). The cues will appear superimposed to a neutral, happy, sad fearful or scrambled face distractors that participant will be told to ignore. Previous studies from our laboratory have demonstrated that without a directional cue, more attentional resources are available to process emotional faces in a goal-directed manner.

The investigators will examine the influence of positive expectations and attention on reaction times and neural processes. Specifically, they hypothesize that older adults will focus more on happy faces and/or less on negative faces compared to neutral faces (i.e. higher/lower reaction times) when more attentional resources are available (attention is not constrained), and that this bias will increase in the positive expectation condition and will be associated with better mood (VAS). Moreover, it is expected that positive expectation effects are related to participants' cognitive control ability. Additionally, the expected positivity and expectation effects will be primarily modulated by the ventromedial prefrontal cortex. This prediction is based on evidence suggesting the preservation of this structure in aging, which compensates for the decline of the dorsolateral prefrontal cortex. Therefore, the investigators predict that positive expectation effects in older adults are related to a shift from the lateral prefrontal cortex to the ventromedial prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 60 years
* MRI compatible
* Medical information and signed declaration of consent
* No history of psychiatric or neurological disorders

Exclusion Criteria:

* Current intake of central nervous system active drugs
* Montreal Cognitive Assessment (MoCA) score below 26
* BMI score above 30
* BDI score above 12

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Effects of positive expectation on mood | Before the intervention (VAS baseline), after 10 minutes, after 25 minutes, after 40 minutes and after the scanning (55 minutes after the baseline) on each day.
  Mood ratings via visual analogue scale (VAS), consisting of a scala from 0 to 400 points (0 meaning unhappy; 400 meaning happy). VAS will be extracted as a raw score and then normalized to the baseline VAS. It will be analyzed following the time course of the experiment and as an average of the VAS measured during the scanner on each day.
Effects of positive expectation on reaction time data | After the intervention, participants will performed this task during 45 minutes while lying in the scanner on each day.
  Reaction times from the emotional interference task will be extracted and sampled for 5 emotional (happy, fearful, sad, neutral and scrambled faces) and 2 attention (high and low attention to faces) conditions and their interaction.
Effects of positive expectation on blood oxygen level dependent (BOLD) signals | Participants will lie in the scanner for approximately 45 minutes while performing the emotional interference task, after the intervention on each day.
  Functional magnetic resonance imaging will be used to extract and analyze BOLD signals (whole brain and regions of interest) in response to the emotional and attention conditions and their interaction.

SECONDARY OUTCOMES:
Fixation and gaze shifts behaviors (eye-tracking) | Participants fixation patterns will be recorded during the performance of the emotional interference task (for 45 minutes) on each day.
  Horizontal gaze trajectories (fixation and gaze shifts patterns) will be recorded using eye-tracking. Data will be extracted and analyzed in degrees of visual angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Systems Neuroscience, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: With publication